CLINICAL TRIAL: NCT00255996
Title: An Open Label Parallel Group Study To Investigate The Pharmacokinetics Of Intravenous Linezolid, An Oxazolidinone, Administered To Healthy Volunteers And Patients With Major Thermal Injuries
Brief Title: Evaluation Of Linezolid Pk Profile In Burns Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5951109
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Linezolid

INTERVENTIONS:
Drug: linezolid

SUMMARY:
Evaluation of linezolid pk profile in burns patients

ELIGIBILITY:
Inclusion Criteria:

* Subject with a Body Mass Index (BMI) < 30 kg/m². For patient with major thermal injuries, the weight will be collected before the burn ;
* Patients with major thermal injuries >40% body area including 3rd degree burns with full thickness burns ;
* Patients hospitalized for at least 10 days since their thermal injury occurred ;

Exclusion Criteria:

* Contra-indications to use linezolid as mentioned in the SmPC (Summarized Product Characteristics) : hypersensitivity to linezolid use or to any of its components, non-controlled hypertension, phaeochromocytoma, carcinoid syndrome, hyperthyroidism, bipolar disorders, schizoaffective disorders, acute confused state of mind, pregnancy, and breastfeeding ;
* Drugs metabolised by monoamine oxydase (MAO) should be evaluated for potential drug-to-drug interaction;
* Subject treated by: selective serotonin reuptake inhibitors (Prozac®, Effexor®, Ixel® …), tricyclic antidepressant (Anafranil®, Sinequan®, Surmontil®, Tofranil®), 5HT1 receptor agonists (triptan) direct or indirect sympathomimetic (including adrenergic bronchodilator, pseudoephedrine and phenylpropylamine), vasopressor (adrenaline and noradrenaline), dopaminergic drugs (dopamine, dobutamine), phenetidine or buspirone should be evaluated for potential drug-to-drug interaction;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To assess and compare pharmacokinetic parameters of a single dose 1-hour intravenous linezolid (Zyvox) at 600 mg in patients with major thermal injuries (>40% body area) and in healthy volunteers

SECONDARY OUTCOMES:
To assess and compare tolerability and safety of a single dose of 600mg IV linezolid administered in patients with major thermal injuries (>40% body area) and in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- France (2):
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951109&StudyName=Evaluation+Of+Linezolid+Pk+Profil+In+Burns+Patients